CLINICAL TRIAL: NCT05663905
Title: A Randomised Controlled Trial to Assess the Efficacy of Intravenous Ambroxol Hydrochloride as an Adjunct Therapy for Severe Pneumonia in Critically Ill Patients
Brief Title: Efficacy of Intravenous Amboxol Hydrochloride as an Adjunct Therapy for Severe Pneumonia in Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JEP-2022-536; FF-2022-376 (Other Grant/Funding Number: Sekretariat Penyelidikan & Inovasi UKM)
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Severe Pneumonia; Community-acquired Pneumonia; Hospital-acquired Pneumonia; Critical Illness
Keywords: mechanical ventilation; severe pneumonia; critical illness; CPIS; Ambroxol
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia; Healthcare-Associated Pneumonia; Critical Illness | interventions — Ambroxol; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ambroxol Arm (Experimental): Amboxol arm will be receiving "standard therapy" as per control group with the addition of IV ambroxol hydrochloride 30mg TDS as adjunct therapy for 14 days. Each dose of 30mg of ambroxol will be diluted in 50ml of NS/D5% to be given intravenously over an hour. The patients will be considered as drop-outs if ambroxol is discontinued due to its side-effects, or if the patient's duration of ICU stay is less than 24 hours.
  Interventions: Drug: Ambroxol Hydrochloride; Other: Standard Therapy
- Control Arm (Other): Control arm will be receiving "standard therapy" for severe pneumonia as per recommended in the ICU Management Protocols by Malaysian Society of Intensive Care (MSIC).37 This includes antibiotics stewardship and supportive therapy.
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Drug: Ambroxol Hydrochloride — IV ambroxol hydrochloride 30mg TDS as adjunct therapy to standard therapy for severe pneumonia in ICU for 14 days. Each dose of 30mg of ambroxol will be diluted in 50ml of NS/D5% to be given intravenously over an hour.
  Other Names: Mucosolvan®; Lasolvan®
  Arms: Ambroxol Arm
Other: Standard Therapy — Standard therapy for severe pneumonia as per recommended in the ICU Management Protocols by Malaysian Society of Intensive Care (MSIC). This includes antibiotics stewardship and supportive therapy.

SUMMARY:
Ambroxol is a mucolytic containing an active N-desmethyl metabolite of bromhexine. It is approved by both the U.S. FDA and EMA to be marketed under several formulations including oral, nasal, oro-mucosal, rectal and intravenous formulations. One of ambroxol's authorized use is for the treatment of bronchopulmonary infections. In addition, it has been found over the decades to have other multi-pronged properties such as local anaesthesia, anti-inflammatory and anti-oxidant effects. It also stimulates surfactant production in Type II pneumocytes, thus preventing atelectasis in pneumonia. Ambroxol has demonstrated a wide safety profile and is an extensively studied drug in terms of safety with the commonest side effects being skin rashes, allergies, nausea, vomiting, abdominal pain and dyspepsia.

Severe pneumonia is is defined by the American Thoracic Society (ATS) as pneumonia that requires ICU admission and specifically fulfils one of two major criteria, or three out of nine minor criteria as per recommended in the latest ATS guideline.

This study aims to investigate the effects of using intravenous ambroxol as an adjunct therapy on the resolution of severe pneumonia. The improvements in modified Clinical Pulmonary Infection Score (CPIS) will be used as a surrogate for resolution of severe pneumonia. Modified CPIS is a clinical score of 0-12 based on 6 clinical features: volume and character of tracheal secretions, chest radiograph infiltrates, body temperature, leukocyte count, oxygenation index, and microbiology results. Traditionally, CPIS score has been used to facilitate the diagnosis of VAP where a cut-off point of >6 is used to denote possible pneumonia. Interestingly, Luna et al has found that serial improvements in CPIS score can be successfully used as a surrogate for pneumonia resolution with good correlation with eventual survivability.

This study will also explore the effects of using ambroxol on other clinical outcomes of patients with severe pneumonia, including ICU mortality, duration of ICU stay, length of mechanical ventilation and incidence of reintubation within 48 hours. If this adjunct treatment is able to reduce duration of ICU stay and length of MV, it will not only directly impact the patients' short & long term outcomes but will also confer logistical benefits in terms of saving resources and reducing healthcare economic burden while optimizing ICU turnover rates.

DETAILED DESCRIPTION:
This prospective, open-label, randomised controlled trial will be conducted in the Intensive Care Unit (ICU) of Universiti Kebangsaan Malaysia Medical Centre (UKMMC). This study protocol will therefore be submitted for the approval of both the Research Committee of Anaesthesiology & Intensive Care Unit, UKKMC and the Research & Ethics Committee of UKMMC prior to its commencement. Written and informed consent will be obtained from the next of kin prior to the commencement of study by the medical doctors in charge of admitting the patients to ICU. These healthcare professionals will be receiving adequate training and information on IV ambroxol hydrochloride and the study protocol in the form of slideshow presentation. The data collection will be done by a single investigator. Intravenous preparation of ambroxol hydrochloride will be imported into Malaysia through customs following the procurement of Clinical Trial Import License.

METHODOLOGY

A total of 32 patients will be recruited based on the inclusion criteria. They will be randomised into either control group (Group C) or intervention group (Group A) using a computer-generated randomiser.

Group C will be receiving "standard therapy" for severe pneumonia as per recommended in the ICU Management Protocols by Malaysian Society of Intensive Care (MSIC). This includes antibiotics stewardship and supportive therapy. Group A will be receiving "standard therapy" as per control group with the addition of IV ambroxol 30mg TDS as adjunct therapy for 14 days. Each dose of 30mg of ambroxol will be diluted in 50ml of NS/D5% to be given intravenously over an hour. The patients will be considered as drop-outs if ambroxol is discontinued due to its side-effects, or if the patient's duration of ICU stay is less than 24 hours.

Data collection will begin from the day of ICU admission until the initial 14 days of ICU stay, until patient is extubated, or death, whichever occurs earlier. Demographic data including age, gender, weight, height, body mass index (BMI), concomitant Covid-19 status and co-morbidities will be documented. Co-morbidities that will be recorded include smoking status, obesity, diabetes mellitus, hypertension, cardiovascular disease, chronic lung disease, chronic kidney disease, malignancy and previous Covid-19 infection.

Clinical data such as ICU admission and discharge date, Acute Physiology and Chronic Health Evaluation II (APACHE II) score on admission, daily Sequential Organ Failure Assessment (SOFA) score, vasopressor requirements, renal replacement therapy during antibiotic therapy, date of intubation and extubation, reason for patient not being extubated by day 14, total duration of mechanical ventilation, incidence of reintubation within 48 hours and ICU outcomes (discharged alive or died in ICU) will also be recorded. The ICU scores used in this study will be used with permission from the publishers of APACHE II and SOFA scores.

Other clinical parameters that will be recorded daily include tracheal aspirate or sputum volume and character, body temperature, leukocyte count, and P/F ratio. Only one data representing the worst value such as highest temperature, lowest PF ratio will be recorded for each parameter daily. Chest X-ray and tracheal aspirate will be taken upon intubation, day 5 and day 10 of treatment. The C-reactive protein and serum procalcitonin level will be taken at less than 3 days and between 5 to 10 days of therapy. Any side effects will be recorded and managed accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years old
* Mechanically ventilated due to severe community or hospital acquired pneumonia

Exclusion Criteria:

* Patients aged <18 years old
* Pregnant and lactating patients
* Patients with known allergies to ambroxol hydrochloride
* Patients with aspartate aminotransferase (AST) >5 times the upper limit of normal at the time of recruitment
* Moribund patients who are expected to not survive within 24 hours of ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Rate of resolution of severe pneumonia | 2 weeks
  Serial CPIS (Clinical Pulmonary Infection Score) will be used to compare rate of resolution of severe pneumonia between the 2 arms

SECONDARY OUTCOMES:
Duration of Mechanical Ventilation | 2 weeks
  Mean duration (in days) of mechanical ventilation between the 2 arms
Length of ICU Stay | 2 weeks
  Mean duration (in days) of ICU stay between the 2 arms
Incidence of ICU mortality | 2 weeks
  Percentage of ICU mortality between the 2 arms will be compared
Incidence of reintubation within 48 hours of extubation | 2 weeks
  Percentage of reintubation within 48 hours of extubation between the 2 arms will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor Dr. Aliza Mohamad Yusof, MD (UKM), Principal Investigator — Hospital Tuanku Muhriz UKM (HCTM)
Locations (1):
- Hospital Canselor Tuanku Muhriz UKM (HCTM), Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No